CLINICAL TRIAL: NCT07101445
Title: Prevent Allergic Reactions to Aphexda With Dexamethasone (PARADE)
Brief Title: Evaluating Premedication Regimens (Methylprednisolone vs Dexamethasone-based) for the Prevention of Systemic and Injection Site Reactions to Motixafortide in Patients With Multiple Myeloma Undergoing Stem Cell Mobilization, PARADE Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Gamida Cell ltd (Industry)
Responsible Party: Principal Investigator, Joseph Cataquiz Rimando, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00008909; NCI-2025-03018 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00008909 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP6478-24 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Acetaminophen; Specimen Handling; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Famotidine; Loratadine; Methylprednisolone; exifone; Medrol Veriderm; montelukast; 4-fluorobenzoyl-TN-14003; BKT140; 4-fluorobenzoyl-Arg-Arg-Nal-Cys-Tyr-Cit-Lys-Lys-Pro-Tyr-Arg-Cit-Cys-Arg-NH2 (S-S bridged); Blood Component Removal; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The labels of the medications will be masked to the patient, the investigator, and the treating nurse.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Dexamethasone) (Active Comparator): See Detailed Description
  Interventions: Drug: Acetaminophen; Procedure: Biospecimen Collection; Drug: Dexamethasone; Other: Electronic Health Record Review; Drug: Famotidine; Drug: Loratadine; Drug: Montelukast; Drug: Motixafortide; Procedure: Pheresis; Other: Questionnaire Administration; Biological: Recombinant Granulocyte Colony-Stimulating Factor
- Arm II (Methylprednisolone) (Experimental): See Detailed Description
  Interventions: Drug: Acetaminophen; Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Drug: Famotidine; Drug: Loratadine; Drug: Methylprednisolone; Drug: Montelukast; Drug: Motixafortide; Procedure: Pheresis; Other: Questionnaire Administration; Biological: Recombinant Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Acetaminophen — Given by mouth (PO).
  Other Names: Acetaminophen (APAP); Paracetamol; Tylenol
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Dexamethasone — Given intravenously (IV).
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Arm I (Dexamethasone)
Other: Electronic Health Record Review — Ancillary studies
Drug: Famotidine — Given by mouth (PO).
  Other Names: Pepcid; Pepcid AC
Drug: Loratadine — Given by mouth (PO).
  Other Names: Claritin
Drug: Methylprednisolone — Given intravenously (IV).
  Other Names: Adlone; Caberdelta M; DepMedalone; Depo Moderin; Depo-Nisolone; Duralone; Emmetipi; Esametone; Firmacort; Medlone 21; Medrate; Medrol; Medrol Veriderm; Medrone; Mega-Star; Meprolone; Methylprednisolonum; Metilbetasone Solubile; Metrocort; Metypresol; Metysolon; Predni-M-Tablinen; Prednilen; Radilem; Sieropresol; Solpredone; Summicort; Urbason; Veriderm Medrol; Wyacort
  Arms: Arm II (Methylprednisolone)
Drug: Montelukast — Given by mouth (PO).
Drug: Motixafortide — Given subcutaneously (SC).
  Other Names: 4F-Benzoyl-TN14003; BKT 140; BKT-140; BKT140; BL 8040; BL-8040; BL8040; TF 14016; TF-14016; TF14016
Procedure: Pheresis — Undergo apheresis
  Other Names: Apheresed; Apheresis; Blood Component Removal; Collection, Apheresis/Leukapheresis; Hemapheresis
Other: Questionnaire Administration — Ancillary studies
Biological: Recombinant Granulocyte Colony-Stimulating Factor — Give Granulocyte Colony-Stimulating Factor (G-CSF).
  Other Names: Recombinant Colony-Stimulating Factor 3; rhG-CSF

SUMMARY:
This phase IV trial compares the effect of premedication regimens with methylprednisolone versus dexamethasone for the prevention of allergic reaction to motixafortide in patients with multiple myeloma (MM) undergoing stem cell mobilization. MM patients that receive an autologous stem cell transplantation (ASCT) have better outcomes. However, not all MM patients are able to have a successful stem cell mobilization and collection which is needed to proceed to ASCT. The addition of motixafortide prior to stem cell mobilization has allowed more MM patients to collect the needed number of stem cells to proceed to ASCT. However, motixafortide does produce systemic and injection site reactions in many patients. The optimal medication regimen to prevent reactions remains unknown. A premedication regimen with dexamethasone prior to motixafortide decreases the incidence of reactions in many patients and is considered the standard of care regimen for the prevention of systemic and injection site reactions to motixafortide in patients with MM undergoing stem cell mobilization. Dexamethasone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen side effects/allergic reactions. However, dexamethasone is associated with other side effects like headache, difficulty sleeping, high blood glucose, high blood pressure, mood changes, fluid retention, and infection, among others. A premedication regimen with methylprednisolone prior to motixafortide may work better to decrease the incidence of reactions to motixafortide in patients with MM undergoing stem cell mobilization. Methylprednisolone is in a class of medications called corticosteroids. It works to decrease side effects/allergic reactions by changing the way the immune system works. Giving methylprednisolone may be safe, tolerable and/or more effective than dexamethasone as part of a premedication regimen for the prevention of allergic reaction to motixafortide in patients with MM undergoing stem cell mobilization.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the safety and efficacy of a premedication regimen for motixafortide that includes loratadine, famotidine, acetaminophen, montelukast, and dexamethasone 12mg intravenously (IV) with an experimental regimen that replaces dexamethasone with methylprednisolone 125mg IV.

SECONDARY OBJECTIVES:

I. Compare the tolerability and patient experience between the regimens. II. Compare the effects of the two regimens on stem cell mobilization. III. Explore the potential immunomodulatory effects of the two regimens.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive granulocyte colony-stimulating factor (G-CSF) once daily (QD) in the morning and loratadine orally (PO) twice daily (BID) on days 1 - 3. Patients receive G-CSF and loratadine PO once in the morning on day 4. Patients then receive loratadine PO, famotidine PO, acetaminophen PO, montelukast PO and dexamethasone IV once in the afternoon on day 4 and 1 hour later receive motixafortide subcutaneously (SC) once in the afternoon on day 4. Patients receive G-CSF once in the morning on day 5 and undergo stem cell apheresis in the morning on day 5. Patients may undergo additional stem cell apheresis on days 6, 7 and/or 8 if target dose of CD34+ cells is not achieved on day 5. Patients may receive additional G-CSF QD in the morning and loratadine PO BID on days 6, 7 and/or 8 if the target dose of CD34+ cells is not achieved on day 5. Patients undergoing additional stem cell apheresis on days 7 and 8 receive loratadine PO, famotidine PO, acetaminophen PO, montelukast PO and dexamethasone IV once in the afternoon on day 6 and 1 hour later receive motixafortide SC once in the afternoon on day 6. Treatment continues in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive G-CSF QD in the morning and loratadine PO BID on days 1 - 3. Patients receive G-CSF and loratadine PO once in the morning on day 4. Patients then receive loratadine PO, famotidine PO, acetaminophen PO, montelukast PO and methylprednisolone IV once in the afternoon on day 4 and 1 hour later receive motixafortide SC once in the afternoon on day 4. Patients receive G-CSF once in the morning on day 5 and undergo stem cell apheresis in the morning on day 5. Patients may undergo additional stem cell apheresis on days 6, 7 and/or 8 if target dose of CD34+ cells is not achieved on day 5. Patients may receive additional G-CSF QD in the morning and loratadine PO BID on days 6, 7 and/or 8 if the target dose of CD34+ cells is not achieved on day 5. Patients undergoing additional stem cell apheresis on days 7 and 8 receive loratadine PO, famotidine PO, acetaminophen PO, montelukast PO and dexamethasone IV once in the afternoon on day 6 and 1 hour later receive motixafortide SC once in the afternoon on day 6. Treatment continues in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo blood sample collection on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged 18 years or older.
* Patient must understand and voluntarily signed an informed consent form.
* Patient must be willing and able to adhere to the study schedule and other protocol requirements.
* Histologically confirmed multiple myeloma prior to enrollment and randomization.
* Eligible for hematopoietic stem cell mobilization and autologous hematopoietic stem cell transplantation as per institutional guidelines.
* Females of reproductive potential must use effective contraception during treatment with motixafortide and for 8 days after the final dose.

Exclusion Criteria:

* Previous history of autologous or allogeneic hematopoietic cell transplantation.
* History of hemoglobin SS disease or hemoglobin S trait precluding the patient's ability to use G-CSF.
* History of steroid-induced psychosis or encephalopathy requiring medical intervention.
* History of type I or II diabetes mellitus that is poorly controlled or with high glucose variability precluding safe administration of dexamethasone 12mg IV as premedication in the opinion of the investigator.
* History of serious systemic reaction to motixafortide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of systemic reactions | At day 4 and 5
  Will compare the incidence and severity of systemic reactions after administration of motixafortide. Systemic reactions will be graded as per Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. Analysis will be based upon an intent-to-treat analysis of all subjects who are randomized to receive dexamethasone or methylprednisolone. Will evaluate the proportion of patients who develop systemic reactions stratified by grade associated with motixafortide between the two premedication regimens. The non-inferiority probability (p)-value between the two arms will be carried out using one-sided z-test. In addition, these two groups will be compared at patient level using chi-square test or Fisher's Exact test. A logistic regression will be used to estimate the odd ratio between the two arms controlling for the baseline covariates for an improved precision of the estimation.
Incidence and severity of injection site reactions | At day 4 and 5
  Will compare the incidence and severity of injection site reactions after administration of motixafortide. Injection site reactions will be graded as per CTCAE v5.0. The incidence of injection site reactions after administration of motixafortide between the two premedication regimens will be similarly compared to that of the incidence and severity of systemic reactions.

SECONDARY OUTCOMES:
Compare Tolerability Between Regimens | At days 4 and 5
  Will compare the change in patient-reported outcomes (PROs) on tolerability before and after administration of the two premedication regimens. Domains will include fatigue, sleep-related disturbances, sleep-related impairment, cognitive function, global functioning, pruritus, and urticaria. Evaluable subjects will be all subjects who were randomized to receive dexamethasone or methylprednisolone. For the (PRO) on tolerability before and after administration of the two premedication regimens, the difference in the mean scores along with the standard deviations for each individual scale (sleep, allergy, injection site reactions and fatigue/function) will be descriptively reported. Internal consistency reliability by Crocbach's alpha for each scale per treatment arm will be evaluated using Crocbach's alpha. Never=1, Rarely=2, Sometimes=3, Often=4, Always=5. Injection Site Reactions Scale: Not at all=1, A little bit=2, Somewhat=3, Quite a bit=4, Very much=5.
CD34+ hematopoietic stem and progenitor cells (HSPC)/kg collection | Up to day 8
  Will compare the median number of CD34+ HSPC/kg collected. Evaluable subjects will be all subjects who were randomized to receive dexamethasone or methylprednisolone. Median number of CD34+ HSPC/kg collected will be compared between the two arms using a Wilcoxon rank-sum test and their respective interquartile ranges will be reported.
Collection of >= 6 x 10^6 CD34+ HSPC/kg | At day 5
  Will compare the number of patients collecting >= 6 x 10^6 CD34+ HSPC/kg within one apheresis procedure. Evaluable subjects will be all subjects who were randomized to receive dexamethasone or methylprednisolone. Comparison between number of patients collecting >= 6 x 10^6 CD34+ HSPC/kg in one apheresis procedure for the two arms will be conducted using the t-test or the Wilcoxon rank-sum test as appropriate.
Cytokine levels | At days 4 and 5
  Will compare the change in plasma cytokine levels before and after administration of the two premedication regimens. Plasma samples for cytokine analysis will be drawn on day 4 prior to premedication administration and then on day 5 prior to apheresis. Cytokine levels will be analyzed by the Winship Cancer Institute core cytokine analysis facilities using multiplex technology. These analyses will focus on Th2 cytokines and mast cell degranulation. Evaluable subjects will be all subjects who were randomized to receive dexamethasone or methylprednisolone. The changes in plasma cytokine levels before and after administration of the two premedication regimens will be descriptively analyzed using means with standard deviations or median with ranges as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rimando, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States